CLINICAL TRIAL: NCT06551662
Title: Drug-coated Balloons vs. Drug Eluting Stents in Bifurcation Coronary Lesions: PICCOLETO V Study
Brief Title: DCB vs. DES in Bifurcation Coronary Lesions
Acronym: PICCOLETO V
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Ricerca e Innovazione Cardiovascolare ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICCOLETO V
Record Dates: First submitted 2024-07-30; First posted 2024-08-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; DCB
Keywords: Coronary artery disease; Bifurcation coronary lesions; Drug-coated balloons
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Device: Paclitaxel drug-coated-balloons (Experimental)
  Interventions: Device: Paclitaxel drug-coated balloons
- Device: Sirolimus drug-coated-balloons (Experimental)
  Interventions: Device: Sirolimus drug-coated balloons
- Device: new generation drug-eluting-stents (Active Comparator)
  Interventions: Device: New generation drug-eluting stent

INTERVENTIONS:
Device: Paclitaxel drug-coated balloons — Patients will be randomized to Paclitaxel drug-coated balloons, Sirolimus drug-coated balloons or standard therapy with new generation drug-eluting stent
  Arms: Device: Paclitaxel drug-coated-balloons
Device: Sirolimus drug-coated balloons — Patients will be randomized to Paclitaxel drug-coated balloons, Sirolimus drug-coated balloons or standard therapy with new generation drug-eluting stent
  Arms: Device: Sirolimus drug-coated-balloons
Device: New generation drug-eluting stent — Patients will be randomized to Paclitaxel drug-coated balloons, Sirolimus drug-coated balloons or standard therapy with new generation drug-eluting stent
  Arms: Device: new generation drug-eluting-stents

SUMMARY:
This is an investigator-driven prospective, multicentric, international, randomized clinical study, in an open-label randomized fashion, where patients with bifurcation coronary artery disease (Medina: 111,101,011,001) in vessels with diameter >2.0 (visual estimation) and with a clinical indication to PCI, will be enrolled. After successful predilatation (with any tool deemed useful), patients will be randomized 1:1:1 to SCB, PCB or standard treatment with DES for bifurcation native vessel disease. All patients with a clinical indication for PCI, both stable coronary artery disease and acute coronary syndrome, will be enrolled.

Before participating all the candidates will be clearly informed about the study, including the possible risks and benefits, and will be asked to provide a written informed consent. Subjects will be instructed that may not meet the general criteria for inclusion or the angiographic criteria, or that may have at least one exclusion criteria, and then be excluded from the study (screening failure), even after informed consent is obtained.

Consecutive patients who meet at least one of the inclusion criteria and none of the exclusion criteria, will participate to the study. After randomization, the procedure will consist in standard coronary angioplasty following international guidelines/consensus documents and as per local practice. If the patient has been randomized to SCB or PCB, it is mandatory to adequately prepare the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be age ≥18 years.
* Subject has silent ischemia, or stable/unstable angina, or acute MI older than 1-week from the onset of chest pain to admission.
* Subject understands the trial design and treatment procedures and provides written informal consent before entering the trial
* Subject is willing to comply with all protocol-required follow-up evaluations.
* Target lesion must be native non-LM bifurcation lesion
* Target lesion must be a bifurcation lesion on coronary angiography (defined as Medina 0,1,1, Medina 1,0,1, Medina 1,1,1 or Medina 0,0,1 coronary bifurcation lesions) and is eligible for percutaneous coronary intervention (PCI).
* Target lesion reference vessel diameter (both main vessel and side branch)

  * 2.0 mm by visual estimation.
* Target lesion must have visually estimated stenosis ≥50%.
* Target lesion length of side branch must be <25 mm by visual estimation.

Exclusion Criteria:

* Patient with STEMI (within 3 days from the onset of chest pain to coronarography).
* Patient has known allergy to the study balloon/stent system.
* Patient has any other serious medical illness that may reduce life expectancy to less than 12 months.
* Patient is pregnant or nursing.
* Patient is participating in another clinical trial that has not reached its primary endpoint within 24 months after the index procedure.
* Patient has a planned procedure that may cause non-compliance with the protocol or confound data interpretation.
* In-stent restenosis lesion.
* Chronic total occlusion (CTO) lesion in either main vessel or side branch.
* Left ventricular ejection fraction <30%;
* Visible and untreatable thrombus at lesion site;
* Target lesion/vessel with any of the following characteristics:

  * Severe and/or >270° calcification of the target vessel, also proximal to the lesion (intravascular imaging);
  * Bifurcation lesion where stent strategy is anticipated;
  * Left main stem stenosis >50%;
  * Target lesion is in the left main stem;
  * Lesions length >50 mm (main vessel)
  * Lesions length >25 mm (side branch)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
6-9 Month CT-FFR or Invasive FFR in Bifurcation Lesions | 6-9-month
  6-9-month CT-scan FFR (core lab)
  * 6-9-month Main vessel CT-FFR
  * 6-9-month Side branch CT-FFR or
  If invasive coronary angiography indicated at 6-9 months:
  * invasive FFR of Main vessel
  * invasive FFR of Side branch
6-9-Month CT-FFR or Invasive FFR: % Max Stenosis (Main + Side Branch) | 6-9-month
  6-9-month CT-scan FFR (core lab):
  * Main vessel % maximum stenosis
  * Side branch % maximum stenosis or
  If invasive coronary angiography indicated at 6-9 months:
  * Main vessel % maximum stenosis
  * Side branch % maximum stenosis

SECONDARY OUTCOMES:
MACE | 24 +/- 1 months
  The MACE was defined as a composite of total mortality, TVR, and spontaneous TV-MI.
Cardiac death | 24+/- 1 months
  Cardiac death rates at 24+/- 1 months follow-up
All-cause death | 24+/- 1 months
  All-cause death rates at 24+/- 1 months follow-up
Q-wave MI | 24+/- 1 months
  Q-wave MI rates at 24+/- 1 months follow-up
Any MI | 24+/- 1 months
  Any MI rates at 24+/- 1 months follow-up
TLR | 24+/- 1 months
  TLR rates at 24+/- 1 months follow-up
TVR | 24+/- 1 months
  TVR rates at 24+/- 1 months follow-up
Vessel thrombosis | 24+/- 1 months
  Vessel thrombosis rates at 24+/- 1 months follow-up
Bleedings following BARC classification | 24+/- 1 months
  Bleedings following BARC classification at 24+/- 1 months follow-up

CONTACTS AND LOCATIONS:
Locations (17):
- Fondazione Ricerca e Innovazione Cardiovascolare, Milan, Italy
- Poland (13):
  - First Department of Cardiology, Medical University of Gdansk, Gdansk, Poland, Gdansk
  - Department of Cardiology and Structural Heart Diseases, Medical University of Silesia, Katowice, Poland, Katowice
  - Department of Interventional Cardiology, Institute of Cardiology, Jagiellonian University Medical College, Kraków, Poland, Krakow
  - Second Department of Cardiology, Jagiellonian University Medical College, Krakow, Poland, Krakow
  - Department of Cardiology, Copper Health Centre (MCZ), Lubin
  - Clinical Department of Interventional Cardiology, Medical University of Lublin, Lublin
  - Department of Cardiology, Poznan University of Medical Sciences, Poznan
  - Department of Cardiology, The Ministry of Internal Affairs and Administration Hospital, Rzeszow, Rzeszów
  - Department of Cardiology and Internal Diseases, Military Institute of Medicine, Warsaw
  - Department of Invasive Cardiology, Centre of Postgraduate Medical Education, Central Clinical Hospital of the Ministry of Interior and Administration, Warsaw
  - Department of Cardiology, Wałbrzych
  - Centre for Heart Disease, University Hospital Wroclaw Department of Heart Disease, Wroclaw Medical University, Wroclaw
  - Third Department of Cardiology, Medical University of Katowice, Zabrze
- Romania (2):
  - Heart Institute, Cluj-Napoca, Cluj-Napoca
  - Sibiu County Emergency Clinical Hospital, Sibiu
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided